CLINICAL TRIAL: NCT02352467
Title: A Multi-Center, Prospective, Randomized Trial Comparing the Effectiveness of Aurix Therapy to Usual and Customary Care in Stage II-IV Pressure Ulcers
Brief Title: Effectiveness of Aurix Therapy in Pressure Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nuo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM004 Gold
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Pressure Ulcer
Keywords: Non Healing Wound
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aurix + UCC (Experimental): Subjects will be treated on average twice a week for the first 2 weeks, and then, once a week thereafter while under active treatment, but actual frequency of treatment will be determined by the treating physician. All subjects will receive Aurix treatment and usual and customary care, which can include advanced therapeutics.
  Interventions: Device: Aurix
- Usual and Customary Care (No Intervention): Subjects will be treated on average twice a week for the first 2 weeks, and then, once a week thereafter while under active treatment, but actual frequency of treatment will be determined by the treating physician. All subjects will receive usual and customary care, which can include advanced therapeutics.

INTERVENTIONS:
Device: Aurix — Aurix is a platelet-rich plasma gel used in the treatment of non-healing wounds. It will be administered twice weekly for 2 weeks then weekly.
  Arms: Aurix + UCC

SUMMARY:
The aim of this trial is to demonstrate the effectiveness of complete wound healing in a prospective, open-label, randomized trial in which pressure ulcers will be treated using Aurix and standard care and compared 1:1 to patients receiving undefined Usual and Customary Care.

DETAILED DESCRIPTION:
Pressure ulcers (PUs) are a common problem in all patient care settings, especially long-term acute care facilities and nursing homes. Aurix is a platelet-rich plasma gel used in the treatment of non-healing chronic wounds. The results of Aurix to date when used to treat PUs have been promising. The aim of this trial is to demonstrate the effectiveness of complete wound healing in a prospective, open-label, randomized trial in which pressure ulcers will be treated using Aurix and standard of care to determine time to heal at 16 weeks. Comparison will be made to patients receiving undefined Usual and Customary Care in a 1:1 manner.

ELIGIBILITY:
Inclusion Criteria:

1. Medicare eligible
2. ≥18 years of age
3. Ulcer of pressure/shear etiology (Stage II, III, and IV, see Appendix 9 for stage definitions)
4. The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (Index Ulcer) that is located on the heel, ischium, sacrum, and trochanter
5. For subjects with potentially multiple eligible PUs, the largest ulcer will be selected as the Index Ulcer for study. There must be at least 4 cm between the Index Ulcer and other ulcers; if all ulcers are closer than 4 cm, the subject should not be enrolled (screen failure)
6. Debrided ulcer size between 3 cm2 and 200 cm2
7. Subject has received UCC care for ≥ 2 weeks at treating wound clinic
8. Demonstrated adequate pressure relief regimen
9. Duration ≥ 1 month at first visit
10. Subject must be willing to comply with the Protocol, which will be assessed by enrolling clinician.

Exclusion Criteria:

1. Subjects known to be sensitive to Aurix components (calcium chloride, thrombin, ascorbic acid) and/or materials of bovine origin
2. Stage I pressure ulcers
3. Ulcers that are unstageable or of deep tissue morphology that have yet to become an open wound
4. Presence of another wound that is concurrently treated and might interfere with treatment of index wound by Aurix
5. Ulcer not of PU pathophysiology (e.g., pure diabetic, vasculitic, radiation, rheumatoid, collagen vascular disease, venous, or arterial etiology)
6. Patients on chemotherapeutic agents or any malignancy in the wound area
7. Subjects who are cognitively impaired
8. Serum albumin of less than 2.5 g/dL
9. Plasma Platelet count of less than 100 x 109/L
10. Hemoglobin of less than 10.5 g/dL
11. Subject has inadequate venous access for repeated blood draw required for Aurix Administration.
12. Life expectancy of < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Time to Heal | 16 weeks
  Compare complete wound healing at 16 weeks for all pressure ulcers treated with Aurix plus standard of care with patients randomized to usual and customary care. Complete wound closure is defined as skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart (FDA Guidance for Industry Chronic Cutaneous Ulcer and Burn Wounds - Developing Products for Treatment, 2006).

SECONDARY OUTCOMES:
Proportion of healed ulcers | 16 weeks
  Proportion of patients with completely healed pressure ulcers
W-QOL (Quality of Life with Chronic Wounds) score | 16 weeks
  Change in mean W-QOL (Quality of Life with Chronic Wounds) score between baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Clausen, PhD, Study Director — Nuo Therapeutics
Locations (22):
- United States (22):
  - Methodist Hospital Wound Care Center, Arcadia, California
  - Beverly Hospital Wound and Hyperbaric Center, Montebello, California
  - Kaweah Delta Rehabiliation Hospital, Visalia, California
  - Bristol Hospital Wound Care Center, Bristol, Connecticut
  - Piedmont, Atlanta, Georgia
  - St. Luke's Wound and Hyperbaric Center, Meridian, Idaho
  - The Center for Wound Healing at FHN, Freeport, Illinois
  - Tufts Medical Center - Center for Wound Healing, Boston, Massachusetts
  - St Joseph Mercy Oakland Hospital Center for Wound Care and Hyperbaric Medicine, Pontiac, Michigan
  - Catskill Regional Medical Center - Wound Healing Center, Harris, New York
  - Orange Regional, Middletown, New York
  - The Wound Center of Niagara, Niagara Falls, New York
  - Onslow Memorial Hospital - Wound Care and Hyperbaric Center, Jacksonville, North Carolina
  - The Center for Wound Healing Crozer Chester Medical Center, Chester, Pennsylvania
  - Aria Health Bucks Wound Center, Langhorne, Pennsylvania
  - Aria Health Frankford Wound Care Center, Philadelphia, Pennsylvania
  - Memorial Hermann Memorial City, Houston, Texas
  - Memorial Hermann South West, Houston, Texas
  - Memorial Hermann South East, Houston, Texas
  - Memorial Hermann Katy Rehab, Katy, Texas
  - St. Mary's Wound and Hyperbaric Center, Huntington, West Virginia
  - The Center for Wound Healing Cabell Huntington Hospital, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No